CLINICAL TRIAL: NCT03630900
Title: 5% O2 or Lower is the Ideal Tension for Culturing Human Embryo Development From Day 3 Onward
Brief Title: Sequential Versus Single O2 Levels on Human Embryo Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banoon IVF Center (Other)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Ibnsina IVF-Oxygen
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Embryo Culture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequential O2 culture (5% then 2.5%) (Experimental): Embryo culture from day 0 to 3 in 5% O2 then split to either 5% or 2.5% O2 until Day 5 or 6.
  Interventions: Other: Sequential O2 Culture
- 5% O2 culture (No Intervention)

INTERVENTIONS:
Other: Sequential O2 Culture — We investigate the effect of sequential O2 levels on human embryo culture after Intracytoplasmic sperm injection (ICSI)
  Arms: Sequential O2 culture (5% then 2.5%)

SUMMARY:
Myriads of elements affect human embryo culture in vitro. These include, but not limited to, air quality, culture media, culture temperature, incubator humidity, pH, and O2 levels. O2 tension has been thoroughly investigated and, to date, 5% O2 level is superior to 20%. Reports showed that lowering the O2 from Day 3 of embryo culture seems to be physiological.

ELIGIBILITY:
Inclusion Criteria:

* ICSI cycles undergoing their first ICSI attempt

Exclusion Criteria:

* ICSI cycles with a previous failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 487 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Ongoing Implantation rate | three months
  number of sacs with a heartbeat after week twelve of gestation

SECONDARY OUTCOMES:
clinical and ongoing pregnancies | three months
  registered pregnancy with fetal heartbeat at week four after transfer and after week twelve of gestation
human embryo development in vitro | three months

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No